CLINICAL TRIAL: NCT01672476
Title: A Randomized, Double-Blind, Multicenter, Phase 3 Study to Evaluate the Antihypertensive Efficacy and Safety of Fimasartan(BR-A-657∙K) 30mg Compared to Placebo in Patients With Mild to Moderate Essential Hypertension
Brief Title: A Multicenter, Phase 3 Study to Evaluate the Antihypertensive Efficacy and Safety of Fimasartan(BR-A-657∙K) 30mg Compared to Placebo in Patients With Mild to Moderate Essential Hypertension
Acronym: fimasartan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Collaborators: Bucheon St. Mary's Hospital (Other); Konyang University Hospital (Other); Korea University Anam Hospital (Other); National Health Insurance Service Ilsan Hospital (Other); Daegu Fatima Hospital (Other); Dong-A University (Other); Soon Chun Hyang University (Other); Asan Medical Center (Other); Gangnam Severance Hospital (Other); Severance Hospital (Other); Ulsan University Hospital (Other); Kangbuk Samsung Hospital (Other); Sejong General Hospital (Other); Ewha Womans University Mokdong Hospital (Other); Jeju National University Hospital (Other); Hallym University Medical Center (Other); Hanyang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A657-BR-CT-L301
Record Dates: First submitted 2012-08-20; First posted 2012-08-27 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Hypertension
Keywords: Fimasartan
MeSH Terms: conditions — Hypertension | interventions — Valsartan; fimasartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): 1 capsule/day of placebo will be orally administered for the study period (8 weeks)
  Interventions: Drug: Placebo
- Valsartan 80mg (Active Comparator): (As reference group) 80mg/day of Valsartan will be orally administered for the study period (8 weeks)
  Interventions: Drug: Valsartan
- Fimasartan 30mg (Experimental): 30mg/day of Fimasartan will be orally administered for the study period (8 weeks)
  Interventions: Drug: Fimasartan

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Valsartan — Valsartan 80mg
  Other Names: Diovan
  Arms: Valsartan 80mg
Drug: Fimasartan — Fimasartan 30mg
  Other Names: Kanarb
  Arms: Fimasartan 30mg

SUMMARY:
A Randomized, Double-Blind, Multicenter, phase III Study to Evaluate the Antihypertensive Efficacy and Safety of Fimasartan (BR-A-657·K) 30mg Compared to Placebo in Patients with Mild to Moderate Essential Hypertension

DETAILED DESCRIPTION:
After subjects have signed informed consent voluntarily, when they are taking hypertension medication, they go through screening period for 7 days including wash-out period.

After screening and wash-out period, subjects take the placebo for 14 days (Maximum 21 days), and evaluate their suitability to Inclusion and Exclusion criteria.

Patients, who evaluated the proper subject for this clinical trial, are allocated to experimental group (Fimasartan 30mg) or Control group (Placebo group) or Reference group (Valsartan 80mg) randomly at a ratio 2:2:1 and their investigational drugs will be administered daily for the study period (8 weeks). Subjects visit their investigators twice during treatment period, when they take their investigational drugs for 4 weeks, and 8 weeks.

The placebo period will be single-blinded and the treatment allocation in this study will be double-blinded.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who agreed to participate in this clinical trial and submitted the written informed consent
2. Subjects aged 20 to 75 years
3. Essential hypertension patients who are measured more 90mmHg, less than 110mmHg of sitting diastolic blood pressure(SiDBP) at baseline(Day 0)
4. Subject who considered to understand this clinical trial, be cooperative,and able to be followed-up whole of the clinical trial period

Exclusion Criteria:

1. Severe hypertension patients: more 110mmHg of mean SiDBP and/or more 185mmHg of mean Sitting systolic blood pressure(SiSBP)
2. Patients with orthostatic hypotension who has sign and symptom
3. Patients with secondary hypertension
4. Patients who are measured the difference of mean blood pressure of one arm under SiDBP 10mmHg or SiSBP 20mmHg at screening and baseline visit
5. Patients who cannot stop administration of hypertension medication through the clinical trial period, and can take any other hypertension medication except investigational drugs
6. Patients with significant investigations-abnormal renal function (Creatinine more 1.5 times than upper limit of normal), abnormal liver function(AST, ALT more 2 times than upper limit of normal), severe fatty liver disease needed medication
7. Patients with clinically significant investigations in laboratory test of screening visit
8. Patients with surgical and medical disease that is able to be affect to absorption, distribution, metabolism and excretion
9. Patients with severe insulin dependent or uncontrolled diabetes mellitus (HbA1c>9, regimen change of oral hypoglycemic agent, using insulin)
10. Patients with severe heart disease, ischemic heart disease within 6 months, peripheral vascular disease, Percutaneous transluminal coronary angiography(PTCA), Coronary artery bypass graft(CABG)
11. Patients with significant ventricular tachycardia, atrial fibrillation, atrial flutter or other significant arrhythmia
12. Patients with hypertrophic obstructive cardiomyopathy, severe obstructive coronary artery disease, aortic stenosis, hemodynamically significant aortic valve or mitral valve disease
13. Patients with severe cerebrovascular disease
14. Patients with wasting disease, autoimmune disease, connective tissue disease at present and/or previous
15. Patients with known severe or malignancy retinopathy
16. Patients with hepatitis B or C or HIV positive reaction
17. Patients with the medical histories of malignant tumor within 5 years,except local basal cell carcinoma of the skin
18. Patients who have a story or evidence of alcohol or drug abuse within 2 years
19. Patients with history of allergic reaction to any angiotensin II antagonist
20. Patients with any chronic inflammation disease needed to chronic inflammation therapy
21. Childbearing and breast-feeding women
22. Female who plan to become pregnancy or have a possibility of pregnancy but don't prevent conception with acknowledged methods
23. Patients who took medicine within 12 weeks from screening visit or is going on the progress of other clinical trial
24. Patients with significant investigations-Hypokalemia(Less than 3.5 mmol/L), Hyperkalemia(exceeded 5.5 mmol/L)
25. Patients with sodium ion or body fluid is deplated and not able to correct
26. Subject who are judged unsuitable to participate in this clinical trial by investigator

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 293 (Actual)
Dates: Start 2012-04; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
the difference of sitting DBP | After 8 weeks from baseline visit
  To compare the difference of sitting DBP between fimasartan 30mg group and placebo group

SECONDARY OUTCOMES:
the difference of sitting DBP | After 8 weeks from baseline visit
  To compare the difference of sitting DBP between fimasartan 30mg group and valsartan 80mg group
the difference of SiDBP | After 4 weeks from baseline visit
  To compare the difference of SiDBP among fimasartan 30mg group, valsartan 80mg and placebo group
the difference of SiSBP | After 4 weeks and 8 weeks from baseline visit
  To compare the difference of SiSBP among fimasartan 30mg group, valsartan 80mg and placebo group
the ratio of responder(SiDBP<90mmHg or ΔSiDBP≥10mmHg) | After 8 weeks from baseline visit
  To compare the ratio of responder(SiDBP<90mmHg or ΔSiDBP≥10mmHg) among fimasartan 30mg group, valsartan 80mg and placebo group
the ratio of subjects who get normalized blood pressure(SiDBP<90mmHg & SiSBP<140mmHg) | After 8 weeks from baseline visit
  To compare the ratio of subjects who get normalized blood pressure(SiDBP<90mmHg & SiSBP<140mmHg) among fimasartan 30mg group, valsartan 80mg and placebo group

CONTACTS AND LOCATIONS:
Overall Officials: Seok Min Kang, M.D., Ph.D., Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Youn JC, Ihm SH, Bae JH, Park SM, Jeon DW, Jung BC, Park TH, Lee NH, Song JM, Yoon YW, Shin ES, Sung KC, Jung IH, Pyun WB, Joo SJ, Park WJ, Shin JH, Kang SM. Efficacy and safety of 30-mg fimasartan for the treatment of patients with mild to moderate hypertension: an 8-week, multicenter, randomized, double-blind, phase III clinical study. Clin Ther. 2014 Oct 1;36(10):1412-21. doi: 10.1016/j.clinthera.2014.07.004. Epub 2014 Aug 3. PMID 25092393